CLINICAL TRIAL: NCT00254982
Title: An Open-Label Study to Determine Equivalence in Efficacy, Organ Safety and Systemic Tolerability Between Infliximab in GROUP I ("High Need") and GROUP II ("Low Need") Patients Suffering From Chronic Plaque Psoriasis (Psoriasis Vulgaris)
Brief Title: Infliximab in High Need Versus Low Need Psoriasis Patients: The IHELP Study (Study P04320)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Essex Pharma GmbH (Industry); Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04320; 2005-001243-28 (EudraCT Number)
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (high-need) (Experimental): Adult participants with moderate to severe plaque psoriasis who were either not controlled by, or were intolerant to or had contraindications to at least two currently available systemic therapies (eg, photochemotherapy, cyclosporine, methotrexate, oral retinoids, fumaric acid esters, efalizumab, etanercept).
  Interventions: Biological: Infliximab
- Group II (low-need) (Experimental): Adult participants with moderate to severe plaque psoriasis who had undergone pretreatment with no more than one currently available systemic therapy (eg, photochemotherapy, cyclosporine, methotrexate, oral retinoids, fumaric acid esters, efalizumab, etanercept).
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab 5 mg/kg was given as an induction regimen at week 0, 2, and 6 weeks after the first infusion and then at week 14.
  Other Names: Remicade; SCH 215596

SUMMARY:
This is an open-label, multicenter, parallel-group comparison study of the efficacy, safety, and tolerability of infliximab therapy in adult patients suffering from chronic plaque psoriasis (psoriasis vulgaris). Patients will be assigned to GROUP I ("high need") or GROUP II ("low-need") by the investigator according to their previous psoriasis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent by the patient for study participation, prior to protocol specific procedures.
* Patients who are 18 years of age or older at time of enrollment, may be male or female and of any race.
* Diagnosis of plaque-type psoriasis (psoriasis vulgaris) at least 6 months prior to screening.
* Plaque-type psoriasis covering at least 10% of total body surface area.
* Psoriasis Area and Severity Index (PASI)-Score of 12 or greater.
* GROUP I ("high need") patients: adult patients with moderate to severe plaque psoriasis who are either not controlled by, or are intolerant to or have contraindications to at least two currently available systemic therapies (e.g. photochemotherapy, cyclosporine, methotrexate, oral retinoids, fumaric acid esters, efalizumab, etanercept). GROUP II ("low need") patients: adult patients with moderate to severe plaque psoriasis who have undergone pre-treatment with no more than one currently available systemic therapy (e.g. photochemotherapy, cyclosporine, methotrexate, oral retinoids, fumaric acid esters, efalizumab, etanercept). A patient showing contraindications towards two systemic treatments, who has never been pretreated with a systemic therapy will be assigned to GROUP II ("low need").
* Patients must have had a chest x-ray (preferably posteroanterior and lateral) within 3 months prior to first infusion with no evidence of malignancy, infection (e.g. tuberculosis) or fibrosis.
* Laboratory test results: liver enzymes (aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transferase (GGT) and alkaline phosphatase) must be within 1.5 times the upper limit of normal range (ULN), total bilirubin <=1.0 ULN, serum creatinine <1.5 mg/dL (must be available at Baseline).
* Patients must agree to avoid prolonged sun exposure or other ultraviolet light sources during the study.
* Women of child-bearing potential must agree to use a medically accepted method of contraception prior to screening, while receiving protocol-specified medication, and for six months after stopping the medication. Acceptable methods of contraception include abstinence, condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device (IUD), oral or injectable hormonal contraceptive, and surgical sterilization (e.g. hysterectomy or tubal ligation).
* Women of child-bearing potential must have a negative serum pregnancy test (beta-human chorionic gonadotropin [hCG]) at Screening (must be available at Baseline).
* Baseline PASI-Score of 12 or greater.

Exclusion Criteria:

* Patients suffering from active or latent tuberculosis. Prior to the start of treatment with infliximab tuberculosis needs to be excluded following the recommendations published by the German Paul Ehrlich Institute.
* Patients who have had or have a serious infection (e.g. abscess, pneumonia or pyelonephritis) or who have been hospitalized or received treatment with intravenous antibiotics during the previous 2 months.
* Patients who are known to be infected with human immunodeficiency virus, hepatitis B or C virus, prior or current opportunistic infections (within the last six months, Herpes zoster within the last 2 months).
* Patients suffering from congestive heart failure including medically controlled asymptomatic patients.
* History of demyelinating disease or symptoms suggestive of multiple sclerosis or optic neuritis.
* Patients who have current signs and symptoms or history of systemic lupus erythematosus.
* Patients suffering from non-plaque psoriasis, e.g. erythrodermic, guttate or pustular forms. The presence of psoriasis-arthritis is no exclusion criterion.
* Patients suffering from current drug induced psoriasis (e.g. a new onset of psoriasis or an exacerbation of psoriasis from beta-blockers or calcium-channel-blockers). If the patient takes one of those substances on a regular basis, it should be on a stable dose for at least three weeks prior to Baseline.
* Patients suffering from severe, progressive or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, cerebral or psychiatric diseases, that, in the opinion of the investigator, would interfere with the study evaluations or safe or optimal participation in the study.
* Any known malignancy during the last five years (except basal cell carcinoma), any history of lymphoproliferative disease.
* Patients who have received any systemic psoriasis therapy (e.g. immunosuppressant) or lithium within 28 days or baseline visit.
* Patients pretreated with etanercept or efalizumab within 28 days of Baseline.
* Patients previously treated with infliximab.
* Patients who have used topical treatments that could affect PASI evaluation (e.g. corticosteroids, anthralin, topical vitamin D derivates) within 2 weeks of baseline visit, except special areas like head or hands.
* Patients who have used any investigational drug within 3 months of Baseline.
* Patients with allergy/sensitivity to study drug or its excipients.
* Women who are breast-feeding, pregnant, or intend to become pregnant.
* Patients with any clinically significant condition or situation, other than the condition being studied.
* Patients who are participating in any other clinical study.
* Patients who are part of the staff personnel directly involved with this study.
* Patients who are a family member of the investigational study staff.
* Patients who have used any investigational drug within 3 months before Baseline.
* Patients who have received any systemic psoriasis therapy (e.g. immunosuppressants) or lithium within 28 days of baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2005-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 (High-need): Adult participants with moderate to severe plaque psoriasis who were either not controlled by, or were intolerant to or had contraindications to at least two currently available systemic therapies (eg, photochemotherapy, cyclosporine, methotrexate, oral retinoids, fumaric acid esters, efalizumab, etanercept). Infliximab 5 mg/kg was given as an induction regimen at week 0, 2, and 6 weeks after the first infusion and then at week 14.
- Group II (Low-need): Adult participants with moderate to severe plaque psoriasis who had undergone pretreatment with no more than one currently available systemic therapy (eg, photochemotherapy, cyclosporine, methotrexate, oral retinoids, fumaric acid esters, efalizumab, etanercept). Infliximab 5 mg/kg was given as an induction regimen at week 0, 2, and 6 weeks after the first infusion and then at week 14.
Period: Overall Study
Arm/Group | Group 1 (High-need) | Group II (Low-need)
Started | 297 | 296
Completed | 261 | 265
Not Completed | 36 | 31
Not completed — Other | 2 | 1
Not completed — Lack of Efficacy | 5 | 3
Not completed — Lost to Follow-up | 5 | 3
Not completed — Adverse Event | 18 | 16
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Inclusion/exclusion criteria violation | 0 | 2
Not completed — Protocol deviation | 1 | 1
Not completed — Diagnosis of Tuberculosis | 1 | 1
Not completed — Malignancy | 0 | 2
Not completed — Opportunistic infection | 1 | 0
Not completed — Abnormal liver function tests | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (High-need) | Group II (Low-need) | Total
Number analyzed (Participants) | 297 | 296 | 593
Age, Customized [Number; unit: Participants]
  <18 years | 0 | 0 | 0
  Between 18 and 83 years | 297 | 296 | 593
  >83 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 101 | 188
  Male | 210 | 195 | 405

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving a Greater Than or Equal to 75% Improvement in Psoriasis Area and Severity Index (PASI75) Score
Description: PASI75 response is defined as participants who achieved at least a 75% improvement in PASI score from Baseline to Week 22. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their responses to therapy. The PASI produces a numeric score that can range from 0 to 72 (the higher the number, the worse the disease).
Time Frame: Baseline and Week 22
Population: Per Protocol Population - All participants in the intent to treat population who completed the study without major protocol violations. For missing data, the last observation carried forward (LOCF) was applied.
Measure: Number; unit: Proportion of participants
Arm/Group | Group 1 (High-need) | Group II (Low-need)
Number analyzed (Participants) | 264 | 265
Proportion of participants | 0.739 | 0.698

ADVERSE EVENTS:
Arm/Group | Group 1 (High-need) | Group 2 (Low-need)
Serious Adverse Events (participants affected / at risk) | 26/297 | 18/296
Other Adverse Events (participants affected / at risk) | 62/297 | 42/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (High-need) (N=297) | Group 2 (Low-need) (N=296)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOVASCULAR DISORDER (Cardiac disorders) | 0 (0) | 1 (1)
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
BLINDNESS UNILATERAL (Eye disorders) | 0 (0) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0)
VITREOUS DISORDER (Eye disorders) | 1 (1) | 0 (0)
DUODENITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2) | 0 (0)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
CHILLS (General disorders) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 3 (3) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 2 (2) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 1 (1)
SUDDEN CARDIAC DEATH (General disorders) | 1 (1) | 0 (0)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1)
SERUM SICKNESS (Immune system disorders) | 2 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WHIPLASH INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 (1) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 3 (3) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LYMPHANGIOSIS CARCINOMATOSA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTATIC RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 1 (1)
EPIDIDYMITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PSORIASIS (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BURSA REMOVAL (Surgical and medical procedures) | 1 (1) | 0 (0)
URETHRAL OPERATION (Surgical and medical procedures) | 0 (0) | 1 (1)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)
SHOCK (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (High-need) (N=297) | Group 2 (Low-need) (N=296)
INFLUENZA LIKE ILLNESS (General disorders) | 20 (22) | 18 (19)
NASOPHARYNGITIS (Infections and infestations) | 30 (35) | 16 (17)
HEADACHE (Nervous system disorders) | 20 (25) | 12 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to pubish or publicly present any interim results of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any elecontronic media) that report any results of study.